CLINICAL TRIAL: NCT03806400
Title: Postoperative Nausea and Vomiting After Paediatric Strabismus Surgery: a Study of Perioperative Modifiable Risk Factors
Brief Title: Postoperative Nausea and Vomit in Strabismus Surgery
Acronym: PONVISS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-204
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Strabismus
Keywords: Postoperative nausea and vomiting; strabismus surgery; oculocardiac reflex
MeSH Terms: conditions — Strabismus; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative nausea and vomiting (PONV) is a major concern in paediatric inpatient surgery and may increase patient discomfort, delay patient discharge, and increase the cost of patient care. The incidence of PONV after strabismus surgery is relatively high, compared with other inpatient surgeries, particularly in children. Oculocardiac reflex (OCR) is a phenomenon defined by bradycardia or dysrhythmia during strabismus surgery. Oculocardiac reflex is commonly caused by the traction on the extraocular muscle (EOM), which, through the ophthalmic branch of trigeminal nerve, stimulates the vagal center. The afferent arm of the reflex is the ophthalmic branch of the trigeminal nerve, and the efferent arm is the vagus nerve, which diminishes sinoatrial node impulses and leads to bradycardia.While there is a general consensus regarding the role of unmodifiable risk factors for PONV, including the number of muscle and the occurrence of Oculocardiac reflex or not, the role of modifiable risk factors, such as duration of surgery and anesthesia and perioperatively administered medications, is still disputed. In the present study, the investigators evaluated whether these factors may be associated with postoperative nausea and vomiting after paediatric strabismus surgery while controlling for a range of covariates.

DETAILED DESCRIPTION:
The primary outcome was incidence of PONV that occurred within 3 days after the operation. The investigators defined PONV as a presence of either nausea or vomiting. In study hospital, it was routine for nurses to assess and record nausea and vomiting every 8 hours for all postoperative patients during postoperative 3 days. Accordingly, the investigators retrospectively collected the presence of PONV from electrical medical records. If patients had discharged hospital within postoperative 3 days, the incidence of PONV was assessed solely during hospital stay. The data, collected included information regarding age at surgery, gender, and type of strabismus. During strabismus surgery, the number and sequence of the operated muscles, HR before traction of the EOM (baseline HR), maximum decreased HR after traction of the EOM, HR at maximum recovery from decreased HR and maintained during traction of the EOM (adrenergic HR), and HR at the cutting of the muscle, were collected. Oculocardiac reflex was defined as a decrease in HR greater than or equal to 20% rather than maximum at first traction of the muscle.

ELIGIBILITY:
Inclusion Criteria:All patients aged from 2-14 years who underwent strabismus surgery under general anesthesia between January 2018 and November 2018 were included in this study. -

Exclusion Criteria:patients with American Society of Anesthesiologists (ASA) physical status III or higher. -

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients aged from 2-14 years who underwent strabismus surgery under general anesthesia between January 2018 and November 2018 were included in this study. -
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | Day 3 postoperative
  Rate of postoperative nausea and vomiting

SECONDARY OUTCOMES:
oculocardiac reflex | through study completion, an average of 1 hour
  Rate of oculocardiac reflex
Number of Participants with operated muscle | through study completion, an average of 1 hour
  Number of Participants with strabismus surgery

OTHER OUTCOMES:
Duration of surgery and anesthesia | through study completion, an average of 1 hour
  Duration of surgery and anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Zhiying Wu, Doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang, China